CLINICAL TRIAL: NCT01749605
Title: A Pilot Comparison of Short-course Nitrofurantoin in Females With Uncomplicated Bacterial Cystitis in the Emergency Department
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Brett A Faine, Clinical Pharmacy Specialist, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201005757
Record Dates: First submitted 2012-12-11; First posted 2012-12-13 (Estimated); Results first posted 2017-04-27 (Actual); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Uncomplicated Bacterial Cystitis
MeSH Terms: interventions — Nitrofurantoin; Ciprofloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- nitrofurantoin 100 mg (Active Comparator)
  Interventions: Drug: Nitrofurantoin monohydrate/macrocrystals 100 mg BID x 3 days
- Ciprofloxacin 250 mg (Active Comparator)
  Interventions: Drug: ciprofloxacin 250 mg BID x 3 days

INTERVENTIONS:
Drug: Nitrofurantoin monohydrate/macrocrystals 100 mg BID x 3 days
  Arms: nitrofurantoin 100 mg
Drug: ciprofloxacin 250 mg BID x 3 days
  Arms: Ciprofloxacin 250 mg

SUMMARY:
Pilot study to compare the efficacy and safety of 3-day, twice-daily regimens of nitrofurantoin and ciprofloxacin in emergency department (ED) patients presenting with UBC.

ELIGIBILITY:
Inclusion Criteria:

* pre-menopausal females
* ages 18-45 years old
* symptoms of a UTI (dysuria, frequency, urgency)

Exclusion Criteria:

* Onset of symptoms >7 days prior to the ED visit
* Non-English speaking
* Symptoms of pyelonephritis
* Diabetic
* Indications of sepsis
* Immunocompromised
* Currently using prophylactic antimicrobials
* Medications that could interfere with study drug
* Pregnant
* Lactating
* History of kidney or liver disease
* Vaginal symptoms
* Presence of a urinary catheter
* Treatment for UBC <2 weeks prior to ED visit
* Known allergy to study drug
* Unavailable for follow-up

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2010-10; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Nitrofurantoin 100 mg: Nitrofurantoin monohydrate/macrocrystals 100 mg BID x 3 days
- Ciprofloxacin 250 mg: ciprofloxacin 250 mg BID x 3 days
Period: Overall Study
Arm/Group | Nitrofurantoin 100 mg | Ciprofloxacin 250 mg
Started | 18 | 17
Completed | 14 | 14
Not Completed | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nitrofurantoin 100 mg | Ciprofloxacin 250 mg | Total
Number analyzed (Participants) | 18 | 17 | 35
Age, Continuous [Mean (Full Range); unit: years] | 24.4 [18 to 44] | 25.1 [18 to 44] | 24.75 [18 to 44]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 17 | 35
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 18 | 17 | 35
Region of Enrollment [Number; unit: participants]
  United States | 18 | 17 | 35

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Cure at Day 7
Description: Seven days after randomization, subjects received a telephone call to determine if their symptoms have completely resolved. Patients answers were limited to: Yes (clinical cure), No (treatment failure)
Time Frame: 7 days
Measure: Number; unit: participants
Arm/Group | Nitrofurantoin 100 mg | Ciprofloxacin 250 mg
Number analyzed (Participants) | 14 | 14
participants | 13 | 12

ADVERSE EVENTS:
Arm/Group | Nitrofurantoin 100 mg | Ciprofloxacin 250 mg
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/17
Other Adverse Events (participants affected / at risk) | 1/18 | 1/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nitrofurantoin 100 mg (N=18) | Ciprofloxacin 250 mg (N=17)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Rash
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) — Nausea and vomiting

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes